CLINICAL TRIAL: NCT06878365
Title: Single-arm Open-label Trial to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BI 3000202 in Adult Patients With Selected Type 1 Interferonopathies
Brief Title: A Study to Test How Well BI 3000202 is Tolerated by People With Type 1 Interferonopathies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1509-0003; 2024-514942-35-00 (Registry Identifier: CTIS); U1111-1309-4909 (Other: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-03-13; First posted 2025-03-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Interferonopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BI 3000202 (Experimental)
  Interventions: Drug: BI 3000202_low dose; Drug: BI 3000202_high dose

INTERVENTIONS:
Drug: BI 3000202_low dose — BI 3000202_low dose
Drug: BI 3000202_high dose — BI 3000202_high dose

SUMMARY:
This study is open to adults with selected type 1 interferonopathies. People can join the study if they have Aicardi-Goutières syndrome (AGS), Coatomer subunit alpha (COPA) syndrome, Familial chilblain lupus (FCL), or another type 1 interferonopathy with a specific gene mutation.

The purpose of this study is to find out how BI 3000202 is tolerated in people with selected type 1 interferonopathies. Participants take a lower dose of BI 3000202 as tablets for 4 weeks. Afterwards, they take a higher dose of BI 3000202 as tablets for 36 weeks. They may continue with the study treatment until every participant has completed 40 weeks of treatment (about 9 months). The participants may also continue their regular treatment for their condition during the study.

During this study, participants visit the study site 13 times or more, depending on when they start their participation. The doctors check the health of the participants and note any health problems that could have been caused by BI 3000202.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients from ≥18 years (or alternative age for adults based on local regulations) to <75 years.
* Genetic diagnosis with mutations in the following affected genes: three prime repair exonuclease 1 (TREX1), ribonuclease H2 subunit A, B or C (RNASEH2B, RNASEH2C, RNASEH2A), SAM And HD domain containing deoxynucleoside triphosphate triphosphohydrolase 1 (SAMHD1), U7 Small Nuclear RNA Associated sm-like protein (LSM11), RNA component of the U7 snRNP (RNU7-1) for AGS; Coatomer subunit alpha (COPA) for COPA syndrome; TREX1, SAM And HD domain containing deoxynucleoside triphosphate triphosphohydrolase 1 (SAMHD1) for Familial chilblain lupus (FCL); DNA nuclease 2 (DNASE2), Adenosine triphosphate synthase family AAA domain containing 3A (ATAD3A) for other type 1 interferonopathies. Genotype documented in medical history is sufficient for eligibility determination and does not require confirmation. Variant identification as "pathogenic" or "likely pathogenic" is preferred according to a joint consensus recommendation of the American College of Medical Genetics and Genomics and the Association for Molecular Pathology. In the absence of such identification, clinical assessment of pathogenicity is required to be documented in the medical records.
* Patients may be either:

  * On standard of care, provided it is on stable doses
  * Not on standard of care
* If women of childbearing potential (WOCBP): must be ready and able to use highly effective methods of birth control. Non-vasectomised male trial participants whose sexual partner is a woman of childbearing potential must be ready and able to use male contraception.

Exclusion Criteria:

* Major chronic inflammatory or connective tissue disease other than selected type 1 interferonopathies, as assessed by the investigator.
* Increased risk of infectious complications based on investigator's judgement.
* Evidence of potential moderate to severe loss of kidney function.
* Evidence of hepatic impairment.
* Further exclusion criteria apply.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-12-06 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse events assessed as related to study drug | Approximately 72 weeks

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 3000202 in plasma from time 0 to 4 hours after administration of the first dose ( AUC0-4) | At Day 1
Maximum measured concentration of BI 3000202 in plasma after administration of the first dose (Cmax) | At Day 1
Area under the concentration-time curve of BI 3000202 in plasma from time 0 to 4 hours at steady state (AUC0-4,ss) | At Days 29 and 85
Maximum measured concentration of BI 3000202 in plasma at steady state (Cmax,ss) | At Days 29 and 85
Predose concentration of BI 3000202 in plasma at steady state immediately before administration of the next dose (Cpre,ss) | At Days 29 and 85
Change from baseline in interferon gene score (IGS) | At baseline, at Week 12

CONTACTS AND LOCATIONS:
Locations (20):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
- Universitair Ziekenhuis Gent, Ghent, Belgium
- France (3):
  - HOP Gui de Chauliac, Montpellier
  - Hôpital Necker, Paris
  - HOP Tenon, Paris
- Germany (3):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Tübingen, Tübingen
- Barzilai Medical Center, Ashkelon, Israel
- Italy (2):
  - ASST degli Spedali Civili di Brescia, Brescia
  - Azienda Sanitaria Universitaria Giuliano Isontina, Trieste
- Portugal (2):
  - ULS de Santa Maria, E.P.E, Lisbon
  - ULS de Santo Antônio, E.P.E - Centro Hospitalar Universitário de Santo António, Porto
- Spain (3):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen del Rocío, Seville
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency